CLINICAL TRIAL: NCT07243717
Title: The Effectiveness of an Information-Assisted Intervention for Potential Living Kidney Donors
Brief Title: Information-Assisted Intervention for Potential Living Kidney Donors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Ching-Hui Chien, RN, PhD, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202102488B0
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Transplant Donation
Keywords: Potential Living Kidney Donors; knowledge; decision self-efficacy; decisional conflict

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Information-Assisted group (Experimental)
  Interventions: Other: Information-Assisted Intervention

INTERVENTIONS:
Other: Information-Assisted Intervention — The intervention content was formulated based on previous Delphi study results and a comprehensive literature review. To facilitate comprehension, the educational materials were presented using illustrations, mind maps, tables, and concise text in an educational manual. Participants may record questions arising during their learning process, which will be discussed and clarified during consultation sessions by members of the transplant team, including physicians, social workers, and transplant coordinators.

SUMMARY:
This study aims to evaluate the effectiveness of an information-assisted intervention in enhancing knowledge, decision self-efficacy, and reducing decisional conflict among potential living kidney donors. Using a one-group pretest-posttest design, participants will be recruited from the urology and kidney transplant outpatient clinics of two hospitals in northern Taiwan. After providing informed consent and completing a baseline questionnaire (T0), participants will receive a four-week information-assisted intervention in addition to routine care, with follow-up assessments at 4 weeks (T1) and 8 weeks (T2). Data will be collected using structured questionnaires assessing decisional conflict, decision self-efficacy, knowledge, positive thinking, family resilience, and satisfaction with the intervention.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of an information-assisted intervention in improving knowledge, decision self-efficacy, and decisional conflict among potential living kidney donors.

A one-group pretest-posttest design will be adopted. During the study period, participants will be recruited through convenience sampling from the urology and kidney transplant outpatient clinics of two hospitals in northern Taiwan. Eligible potential donors who have completed medical examinations and return for follow-up visits to review tissue matching and laboratory test results will be invited to participate in the study (experimental group). After providing informed consent, participants will complete a baseline questionnaire (T0) in a private setting.

Participants will then receive the information-assisted intervention, followed by the first posttest (T1) at 4 weeks and the second posttest (T2) at 8 weeks after T0. In addition to routine care, the experimental group will receive a four-week information-assisted intervention.

Data will be collected using structured questionnaires, including the Decisional Conflict Scale, Decision Self-Efficacy Scale, Knowledge Test on Living Kidney Donation, Demographic and Clinical Characteristics Questionnaire, Positive Thinking Scale, Evaluation Form for the Information-Assisted Program, and the Family Resilience Scale.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo evaluation for living kidney donation
* Owns a smartphone or tablet with internet access
* Able and willing to participate in the study and provide written informed consent

Exclusion Criteria:

- Deemed unsuitable for kidney donation after evaluation by a transplant specialist

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Decision Self-Efficacy Scale | Baseline (T0, prior to intervention), 4 weeks (T1) and 8 weeks (T2) after Baseline
  The Chinese version of the Decision Self-Efficacy Scale from the Ottawa Hospital Research Institute will be used. This 11-item scale measures individuals' confidence in making informed decisions. Each item is scored from 0-4, with total scores converted to a range of 0-100. Higher scores reflect stronger decision self-efficacy.
Decisional Conflict Scale | Baseline (T0, prior to intervention), 4 weeks (T1) and 8 weeks (T2) after Baseline
  The study will employ the Chinese version of the Decisional Conflict Scale developed by the Ottawa Hospital Research Institute. The 16-item scale uses a 0-4 rating system (0 = yes, 4 = no). Total scores are calculated as (sum of items ÷ number of items) × 25, yielding a range of 0-100. Higher scores indicate greater decisional conflict.
Knowledge Test on Living Kidney Donation | Baseline (T0, prior to intervention), 4 weeks (T1) and 8 weeks (T2) after Baseline
  A 31-item self-developed test will assess participants' knowledge regarding living kidney donation, including anatomy, legal regulations, donor eligibility, medical coverage, surgical risks, postoperative complications, and post-surgical care. Each question has three options: True, False, and Unclear. Correct answers receive 1 point, while incorrect or unclear answers receive 0 points. Higher total scores indicate better knowledge.

SECONDARY OUTCOMES:
Positive Thinking Scale | Baseline (T0, prior to intervention), 4 weeks (T1) and 8 weeks (T2) after Baseline
  The Chinese version of the Positive Thinking Scale will be employed to assess participants' optimism and goal orientation. The 18-item instrument has a total score range of 18-80, where higher scores indicate greater personal satisfaction and goal pursuit.

OTHER OUTCOMES:
Family Resilience Scale | Baseline (T0, prior to intervention)
  The Short Form of the Chinese Family Resilience Assessment Scale (FRAS) will be used to measure family resilience among potential donors. Each of the 32 items is rated on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree), producing total scores from 32 to 128. Higher scores reflect greater family resilience.
Evaluation of the Information-Assisted Program | 4 weeks (T1) after Baseline
  A five-item self-developed questionnaire will be used to evaluate participants' acceptance and satisfaction with the intervention. Scores range from 0-100, with higher values indicating stronger satisfaction and agreement that the intervention was beneficial and appropriate for future potential donors.
Demographic and Clinical Characteristics-Age | Baseline (T0, prior to intervention)
  Actual age (years)
Demographic and Clinical Characteristics-Sex | Baseline (T0, prior to intervention)
  Male / Female
Demographic and Clinical Characteristics-Marital Status | Baseline (T0, prior to intervention)
  Single, Married, Divorced, Separated, Widowed, Cohabiting
Demographic and Clinical Characteristics-Education | Baseline (T0, prior to intervention)
  None, Elementary, Junior High, Senior High, College/University, Graduate/Doctorate, Other
Demographic and Clinical Characteristics-Religion | Baseline (T0, prior to intervention)
  None, Taoism, Buddhism, Catholicism, Christianity, I-Kuan Tao, Other
Demographic and Clinical Characteristics-Occupation | Baseline (T0, prior to intervention)
  None, Physically demanding, Mentally demanding, Both, Neither, Retired, Other
Demographic and Clinical Characteristics-Relationship to Recipient | Baseline (T0, prior to intervention)
  Spouse, Sibling, Parent-child, Relative, Other
Demographic and Clinical Characteristics-Perceived Health Status | Baseline (T0, prior to intervention)
  One item; Score range 0-100; higher = better health perception
Demographic and Clinical Characteristics-Chronic Diseases | Baseline (T0, prior to intervention)
  None, Diabetes, Hypertension, Heart disease, Asthma, Bronchitis, Other
Demographic and Clinical Characteristics-Serum Creatinine (mg/dL) | Baseline (T0, prior to intervention)
  Higher values indicate poorer renal function
Demographic and Clinical Characteristics-24-h Creatinine Clearance (mL/min) | Baseline (T0, prior to intervention)
  Higher values indicate better renal function
Demographic and Clinical Characteristics-Estimated GFR (mL/min/1.73m²) | Baseline (T0, prior to intervention)
  Higher values indicate better renal function
Demographic and Clinical Characteristics-Urine Protein | Baseline (T0, prior to intervention)
  None, Present, Other
Demographic and Clinical Characteristics-Serum Creatinine-Body Weight (kilograms) | Baseline (T0, prior to intervention)
  Measured in kilograms
Demographic and Clinical Characteristics-Height (centimeters) | Baseline (T0, prior to intervention)
  Measured in centimeters
Demographic and Clinical Characteristics-Information Source | Baseline (T0, prior to intervention)
  None, Physician, Transplant Coordinator, Nurse/NP, Other
Demographic and Clinical Characteristics-Decision Status | Baseline (T0, prior to intervention), 4 weeks (T1) and 8 weeks (T2) after Baseline
  No, Considering, Yes
Demographic and Clinical Characteristics-Family Support | Baseline (T0, prior to intervention)
  Supportive, Neutral, Not supportive
Recipient-Related Clinical Data-Dialysis Treatment | Baseline (T0, prior to intervention)
  Yes / No (Hemodialysis or Peritoneal Dialysis)
Recipient-Related Clinical Data-Serum Creatinine (mg/dL) | Baseline (T0, prior to intervention)
  Higher values indicate poorer renal function

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data supporting this study's findings are available from the corresponding author upon reasonable request. The data are not publicly available due to the consideration of ethics, the researchers shall maintain the privacy of the participants, and research data should be used only for academic articles.